CLINICAL TRIAL: NCT03303573
Title: Safety and Efficacy of Repetitive Erythropoietin Treatment for Cerebral Palsy
Brief Title: Safety and Efficacy of Multiple EPO Injections in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, M.D., Professor, Bundang CHA Hospital
Other Study IDs: Multiple EPO
Record Dates: First submitted 2017-08-18; First posted 2017-10-06 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Palsy
Keywords: Erythropoeitin
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- recombinant human erythropoietin group: cerebral palsy patients who had received erythropoietin from January 2013 to November 2016
  Interventions: Drug: recombinant human erythropoietin

INTERVENTIONS:
Drug: recombinant human erythropoietin — Subcutaneous rhEPO injection
  Other Names: rhEPO

SUMMARY:
This study is a retrospective review on the safety and efficacy of repetitive erythropoietin injection in children with cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy is mostly caused by hypoxic-ischemic encephalopathy from preterm birth, involving inflammatory and apoptotic cellular response. Erythropoietin (EPO) has shown neuroprotective effects via activation of anti-inflammatory, angiogenic, and anti-apoptotic pathways. The safety and feasibility of EPO in children were proven in previous clinical trials. In addition, the efficacy of EPO is actively being investigated and some reports have shown potential benefits in cerebral palsy. To confirm the safety and efficacy of multiple injections with expected effect, retrospective review on medical records was performed.

ELIGIBILITY:
Inclusion Criteria:

* confirmed clinical diagnosis of cerebral palsy based on neuromotor findings,
* less than 18 years of age,
* received recombinant human erythropoietin (rhEPO) more than once.

Exclusion Criteria:

* not responding to phone interview or
* no functional assessments available.

Age Groups: Child, Adult, Older Adult
Study Population: Children diagnosed with cerebral palsy who had received recombinant human erythropoietin more than once.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | interview was performed at an average of 1 year after the completion of rhEPO injections
  telephone interview was conducted to collect information of adverse events from all patients.

SECONDARY OUTCOMES:
Change of Gross Motor Function Measure | The results between the baseline evaluation before rhEPO injection and the last evaluation at an average of 1 year after rhEPO injections were compared
  The change of GMFM score before and after rhEPO injections

IPD SHARING:
Plan to Share IPD: Undecided